CLINICAL TRIAL: NCT05139277
Title: Clinical Investigation to Evaluate the CONVIVO System for Discrimination of Normal From Abnormal Tissue During Brain Tumor Resection
Brief Title: Evaluation of the CONVIVO System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Principal Investigator, Linton T. Evans, Principle Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D20056; NCI-2023-06342 (Other: National Cancer Institute)
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma; Glial Tumor; Brain Metastases; Meningioma; Schwannoma; Pituitary Tumor
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms; Meningioma; Neurilemmoma; Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: Adult patients (age>18) presenting with suspected intracranial gliomas (including glioblastoma), cerebral metastasis, meningiomas, acoustic neuromas, and pituitary adenomas, who are surgical candidates and provide informed consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CONVIVO system (Experimental): During tumor resection, study investigators trained in the use of the system will determine when the CONVIVO imaging system will be used for in vivo¬ imaging. At this point 5 mg/kg of fluorescein will be administered intravenously by an anesthesia provider over one minute.Approximately 2-5 minutes following administration of FNa in situ imaging will be performed by the participating surgeon ensuring proper technique.
  Interventions: Diagnostic Test: CONVIVO system
- Conventional histologic evaluation (Other): Following image acquisition, the tissue region imaged with the CONVIVO system will then be biopsied using biopsy forceps. This will be passed immediately off the surgical field as a research specimen and provided to a member of the research team to be prepared for conventional histologic evaluation. The specimen will be labeled with the deidentified subject and sample number. This sequence will then be repeated for each successive sample.
  Interventions: Other: Conventional histologic evaluation

INTERVENTIONS:
Diagnostic Test: CONVIVO system — Approximately 2-5 minutes following administration of FNa in situ imaging will be performed by the participating surgeon ensuring proper technique. Prior to entering the surgical field, the probe will be covered in a disposable sterile sheath that is manufactured with quality assurance for this purpose. The probe will gently be held against the tissue interface while imaging occurs. Again this will only be in regions that would normally be resected or sampled in routine clinical care. Following image acquisition, a neuropathologist present in the operating room, will review and capture each image.
  Arms: CONVIVO system
Other: Conventional histologic evaluation — Following image acquisition, the tissue region imaged with the CONVIVO system will then be biopsied using biopsy forceps. This will be passed immediately off the surgical field as a research specimen and provided to a member of the research team to be prepared for conventional histologic evaluation. The specimen will be labeled with the deidentified subject and sample number. This sequence will then be repeated for each successive sample.
  Arms: Conventional histologic evaluation

SUMMARY:
The primary objective of this study is to evaluate the diagnostic performance of the CONVIVO confocal endomicroscope in discriminating between normal and abnormal tissue in vivo during brain tumor surgery. The interpretation of intraoperative images obtained in situ will be tested against conventional histologic evaluation of targeted biopsies from imaged tissue. The study team hypothesize that there will be a high degree of correlation between images obtained with the CONVIVO system and conventional histologic interpretation.

DETAILED DESCRIPTION:
The surgical resection of brain tumors is an integral component of modern neuro-oncology. . Extent of resection has been found to be associated with increased overall and progression free survival, with the greatest benefit occurring in the setting of a complete or gross total resection. Unfortunately, there are a number of obstacles unique to brain tumors that may limit the extent of resection. A number of advancements in neurosurgical oncology have emerged to improve the extent of tumor resection while decreasing operative morbidity and mortality. Confocal reflectance microscopy is a routine technique used to visualize tissues without fixation or staining used in classical histological techniques. Laser scanning confocal microscopy (LSCM) is an optical fluorescence imaging modality used for imaging thick in vivo and ex vivo tissues. Clinically available confocal endomicroscopy systems contain lasers with precise excitation wavelengths and dichroic filters for detecting appropriate emission wave lengths. The studies completed to date do not evaluate the ability of confocal microscopy to discriminate between normal and abnormal tissue at the margins during surgical resection. This is the first of such in vivo feasibility studies that aims to demonstrate this claim of the CONVIVO system.

The images acquired with the CONVIVO system following administration of fluorescein will be compared to conventional histologic specimens from corresponding biopsies. This is a planned single center study. This study is designed to assess the diagnostic accuracy of the CONVIVO system compared with gold-standard histopathology in tissue that has already been identified for resection. The device will not be used to inform surgical decision making, nor will tissue that would not otherwise be resected be biopsied for research purposes.

This study will rely on study investigators, all physicians at Dartmouth-Hitchcock, to identify subjects. Written consent is required for participation in the study.. There are no specific medical risks to patients associated with the use of CONVIVO. It is not anticipated that there are immediate or direct benefits to patients participating in this study. The CONVIVO imaging data acquired during the procedure will be initially stored on the device's hard drive and later securely uploaded to an encrypted Dartmouth-Hitchcock server. Patients will have the ability to maintain their privacy with minimal disruption or contact by the study team. Additionally, the PI or other investigators will have interactions with the patient as part of their routine clinical care. Participants are free to withdraw from participation in the study at any time upon request.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age>18)
* Adults presenting with suspected intracranial gliomas (including glioblastoma), cerebral metastasis, meningiomas, acoustic neuromas, and pituitary adenomas, who are surgical candidates
* Adults able to provide informed consent.

Exclusion Criteria:

* Pregnancy
* Children (age <18 years)
* Fluorescein sodium (FNa) allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of CONVIVO in discriminating between normal and abnormal tissue | On day of Surgery, Day 0
  Concordance between in vivo imaging with the CONVIVO system and conventional histologic assessment.The diagnostic performance of the CONVIVO system will be assessed with respect to classification as "normal" or "abnormal" tissue. The interpretation of intraoperative images obtained in situ will be tested against conventional histologic evaluation of targeted biopsies from imaged tissue. Pertinent tumors include all intracranial neoplasms including low and high grade glial neoplasms, glioneuronal tumors, cerebral metastasis, meningioma, schwannoma, and pituitary lesions.

SECONDARY OUTCOMES:
Degree of concordance with histologic diagnosis | On day of surgery, Day 0
  Degree of concordance between in vivo imaging with the CONVIVO system and conventional histologic assessment or frozen with respect to histologic diagnosis.
Sensitivity and Specificity of CONVIVO system | On day of surgery, Day 0
  Sensitivity and specificity analysis of CONVIVO using area under the curve and receiver operating characteristics. Conventional histopathology will be the gold-standard.
Rate of uninterpretable or non-diagnostic imaging with the CONVIVO system. | On day of surgery, Day 0
  Rate of uninterpretable or non-diagnostic imaging with the CONVIVO system. During the resection the PI or other investigators may image tissue that is ultimately not biopsied. For example at the end of resection if there is a region of interest that cannot be safely resected, the CONVIVO system can be used to image the tissue without obtaining a corresponding tissue specimen for histology. During image acquisition it will be noted and documented by the research team that there is not a corresponding tissue specimen.
Correlation between intra-operative confocal microscopy and co-registered MRI points. | On day of surgery, Day 0
  MRI characteristics will include (i) the presence or absence of contrast enhancement; (ii) signal intensity on T2 weighted images; (iii) perfusion based and spectroscopy imaging; (iv) diffusion weighted sequences.
Correlation between visible yellow-light fluorescence (560 nm filter) and intraoperative confocal microscopy. | On day of surgery, Day 0
  Following image coregistration, the 560 yellow light filter on the Kinevo microscope will be used to determine the visible fluorescence in the region that was interrogated and classified from 0 to 4 based upon the fluorescence intensity. This will be recorded by the research team. The degree of visible fluorescence will be graded as 0-no fluorescence, 1- weak intensity, 2-moderate intensity, 3-strong intensity.
Correlation between visible blue-light fluorescence and quantitative fluorescence measurements | On day of surgery, Day 0
  If the participant has also received 5-ALA, the 400 nm blue light filter will then be selected and the visible fluorescence of PPIX will also be classified from 0 to 4 based upon the fluorescence intensity. The degree of visible fluorescence will be graded as 0-no fluorescence, 1- weak intensity, 2- moderate intensity, 3-strong intensity.
Extent of tumor resection | 2 Days after surgery up to one month.
  Extent of resection has been found to be associated with increased overall and progression free survival, with the greatest benefit occurring in the setting of a complete or gross total resection. Postoperative MRI is obtained as appropriate, as it relates to extent of resection.
Adverse events related to the administration of fluorescein | Day of surgery (Day 0), 2 Days after surgery up to one month.
  Record adverse events as reported by participant or observed by investigator related to the administration of fluorescein
Time to interpretation of imaging and histology | Day of surgery (Day 0), and up to one week
  Time to pathologic interpretation of intraoperative imaging compared to conventional interpretation of histology.Currently, the frozen section provides intraoperative histopathological analysis of brain tumors. Though useful, this process is time consuming and requires the cutting, freezing, and staining of several biopsies.
Ability to discriminate between viable tumor and pseudoprogression or "treatment effect" using the CONVIVO system. | Day of surgery (Day 0) and up to one month
  The WHO criteria for the diagnosis of Glioblastoma (GBM) - cell density, cellular pleomorphism, increased mitoses, microvascular proliferation and trpalisading or ischemic necrosis - were all detectable by Confocal EndoMicroscope (CEM). Identification of the infiltration zone or the center of the tumor was possible based upon assessments of cell density comparing the center and border specimens. Additional aspects, e.g. apoptotic figures in perinecrotic pseudopalisading tumor cells, and important histological structures such as giant cells, fibrillary tumor matrix and blood vessels were also visible with CEM. Typical features of CEM in patients with histologically proven meningioma were also seen.

CONTACTS AND LOCATIONS:
Overall Officials: Linton T Evans, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans at this time to share IPD.